CLINICAL TRIAL: NCT03505996
Title: A Single-Arm, Multicenter, Phase II Clinical Trial of CS1001 in Subjects With Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: A Study of CS1001 in Subjects With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1001-202; CTR20180423 (Registry Identifier: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2018-04-15; First posted 2018-04-23 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS1001 (Experimental): Participants will receive CS1001 1200 mg by intravenous infusion every three weeks
  Interventions: Biological: CS1001

INTERVENTIONS:
Biological: CS1001 — Monoclonal antibody

SUMMARY:
This is a multicenter, single-arm phase II study to evaluate the efficacy and safety of CS1001 monotherapy for relapsed/refractory classical Hodgkin Lymphoma (rr-cHL)

DETAILED DESCRIPTION:
Eligible subjects with rr-cHL who failed at least two prior lines of therapies are planned to receive CS1001 1200 mg intravenous infusion every three weeks until progression of disease, intolerable toxicity, consent withdrawn or death.The primary endpoint of this trial is objective response rate (ORR), as assessed by independent radiological review committee (IRRC) based on Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically confirmed cHL at study site.
2. Relapsed or refractory cHL that failed at least two lines of systemic therapy.
3. ECOG PS of 0-2.
4. Subjects with at least one measurable lesion at baseline.
5. Subjects treated by prior anti-cancer therapy whose toxicity resolved to baseline or =< Grade 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03
6. Subjects who agree to use highly effective contraception.

Exclusion Criteria:

1. Nodular lymphocyte predominant Hodgkin lymphoma or grey zone lymphoma.
2. Primary site in central nervous system (CNS) or CNS involvement.
3. Subjects currently participating in other clinical studies or use of any investigational drug within 4 weeks prior to the first dose of CS1001.
4. Subjects who had systemic corticosteroid or any other immunosuppressive therapy within 14 days prior to the first dose of CS1001.
5. Subject who had chemotherapy, immune therapy or biological therapy as systemic anti-cancer treatment within 28 days prior to the first dose of CS1001.
6. Receipt of traditional medicinal herbal preparations within 7 days prior to the first dose of CS1001.
7. Known history of human immunodefiency virus (HIV) infection and/or acquired immune deficiency syndrome.
8. Subjects with active Hepatitis B or C infection.
9. Subjects with active tuberculosis infection.
10. Subjects who received prior therapy with anti-PD-1, anti-PD-L1 or anti CTLA-4 monoclonal antibody.
11. Female subjects who are pregnant or breast-feeding.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From first patient first visit to 6 month after last patient first visit
  The percentage of subjects whose best overall response is either complete response or partial response evaluated by IRRC according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China